CLINICAL TRIAL: NCT06205485
Title: A Phase 3 Randomized Trial Of Neoadjuvant Chemotherapy, Excision And Observation Versus Chemoradiotherapy For Early Rectal Cancer
Brief Title: Neoadjuvant Chemotherapy, Excision And Observation vs Chemoradiotherapy For Rectal Cancer
Acronym: NEO-RT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Alliance for Clinical Trials in Oncology (Other); ECOG-ACRIN Cancer Research Group (Network); NRG Oncology (Other); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTG-CO32; CCTG-CO32 (Other: NCI/CTEP); NCI-2023-10515 (Other: NCI CTRP)
Record Dates: First submitted 2023-12-11; First posted 2024-01-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Leucovorin; Oxaliplatin; Fluorouracil; Capecitabine; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- FOLFOX OR CAPOX (Active Comparator): FOLFOX= Six cycles of modified FOLFOX consisting of leucovorin, oxaliplatin and bolus fluoruracil (optional), infusional fluorouracil.
  CAPOX= Capecitabine twice daily for 14 days and Oxaliplatin on day 1
  Interventions: Drug: Leucovorin; Drug: Oxaliplatin; Drug: Fluoruracil; Drug: Capecitabine
- ChemoRT (Active Comparator): Standard dose of infusional 5-Fluorouracil/capecitabine and radiation
  Interventions: Drug: Fluoruracil; Drug: Capecitabine; Radiation: Radiation

INTERVENTIONS:
Drug: Leucovorin — 400 mg/m2
  Arms: FOLFOX OR CAPOX
Drug: Oxaliplatin — 85 mg/m2 or 130 mg/m2 on day 1
  Arms: FOLFOX OR CAPOX
Drug: Fluoruracil — bolus fluoruracil (optional) 400 mg, infusional fluorouracil 2,400 mg/m2
Drug: Capecitabine — 1,000 mg/m2 twice daily for 14 days
Radiation: Radiation — 54 Gy (27-30 fractions)
  Arms: ChemoRT

SUMMARY:
This study is being done to answer the following questions: Is the chance of rectal cancer responding the same if chemotherapy alone is given before limited surgery compared to chemotherapy and radiation therapy given together before limited surgery? If radiation therapy is not given, is quality of life better?

DETAILED DESCRIPTION:
This study is being done to find out if this approach is better or worse than the usual approach for early rectal cancer. The usual approach is defined as care most people get for early rectal cancer.

The usual approach for patients who are not in a study is surgery to remove the rectum or treatment with chemotherapy and radiation therapy, followed by surgery. There are several chemotherapy drugs approved by Health Canada that are commonly used with radiation therapy. For patients who get the usual approach for this cancer, about 90 out of 100 are free of cancer after 5 years.

If a patient decides to take part in this study, they will either get a combination of chemotherapy drugs called FOLFOX or CAPOX for up to 12 weeks or will get chemotherapy with radiation therapy for up to 6 weeks.

After finishing treatment, and even if treatment is stopped early, the study doctor will watch for side effects and determine which type of surgery would be best. After surgery, patients will be asked to come in every 4 months for 2 years, then every 6 months for an additional year. Then will be checked every year for 2 years. This means seeing the study doctor for up to 5 years after surgery. Patients may be seen more often if your study doctor thinks it is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive, well-moderately differentiated rectal adenocarcinoma, mismatch repair proficient.
* MRI stage cT1 not eligible for transanal surgery or cT2-T3ab*. * T3a: <1mm depth invasion, T3b: 1-5mm depth of invasion.
* cN0 stage based on pelvic MRI - including absence of radiographic evidence of mesorectal nodal metastasis, tumour deposits or extramural venous invasion (EMVI).
* M0 stage based on no evidence of metastatic disease by CT imaging of chest, abdomen and pelvis.
* Mid to low-lying tumour eligible for transanal excision in the opinion of the treating surgeon.
* Medically fit to undergo radical TME surgery as per treating surgeon's decision.
* Participant is able (i.e. sufficiently fluent) and willing to complete the quality of life questionnaires in either English or French or Spanish.
* Age of at least 18 years.
* No contraindications to protocol chemotherapy.
* Adequate normal organ and marrow function: ANC ≥ x 10^9/L; platelet count ≥ 100 x 10^9/L; bilirubin < 1.5 UNL, excluding Gilbert's syndrome; Estimated creatinine clearance of ≥ 50ml/min
* Patient must have an ECOG performance of <2 (or Karnofsty ≥ 60%).
* Must be accessible for treatment and follow-up
* Males and females of reproductive potential must have agreed to use a highly effective contraceptive method during and for 6 months after completion of chemotherapy.
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.

Exclusion Criteria:

* Pathologic high-risk factors on diagnostic biopsy: high histologic grade (poorly differentiated), mucinous or signet ring histology.
* Patients with visible pelvic sidewall nodes on MRI.
* Patients with unequivocal determination of nodal disease that, in the opinion of the investigator, would prohibit protocol therapy administration.
* Previous pelvic radiation for any reason, including brachytherapy alone.
* Patients who have had primary lesion excised prior to enrollment. If a patient has had partial excision prior to enrollment, there must be gross residual disease endoscopically for patient to be eligible.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Prior treatment for rectal cancer.
* Patients with known dihydropyrimidine dehydrogenase deficiency (DYPD).
* Potential trial participants should have recovered from clinically significant adverse events of their most recent therapy/intervention prior to enrollment.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Any contra-indications to undergo MRI imaging.
* Presence of anterior lesions above or near peritoneal reflection rendering the patient ineligible for a transanal tumour excision.
* T3 tumours invading or abutting the internal sphincter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2030-01-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate upon re-staging | 6 years
Quality of Life defined using the LARS score | 6 years

SECONDARY OUTCOMES:
Total Mesorectal Excision (TME) Free Survival | 6 years
  Defined as time from randomization to the time of TME attempt or performance, local recurrence after complete clinical response (cCR), or death from any cause
Disease Free Survival | 6 years
  Defined as time from randomization to local recurrence/regrowth after cCR that cannot be salvaged with an R0 TM, M1 recurrence, or death
Overall Survival | 6 years
  Among patients treated with induction chemotherapy versus chemoradiotherapy
Rate of downstaging to ypTO/1N0/X | 6 years
Bowel function assessed by Low Anterior Resection Syndrome (LARS) Score | 6 years
Bladder function assessed by EORTC QLQ-CR29 urinary frequency and urinary incontinence subscales | 6 years
Other QoL functions assessed by subscales of FIQL | 6 years
Other QoL functions assessed by subscales of EORTC QLQ-C30 | 6 years
Other QoL functions assessed by subscales of subscales of EORTC QLQ-CR29 | 6 years
Number and severity of adverse events utilizing CTCAE v5.0 | 6 years
Validate the magnetic resonance tumour regression grade (MR-TRG) in patients with T1-T3a rectal cancer | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Kennecke, Study Chair — Providence Portland Medical Centre, Portland, OR, USA; Carl Brown, Study Chair — St. Paul's Hospital, Vancouver, BC, Canada
Locations (100):
- United States (95):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Rush-Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - The Community Hospital, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - East Carolina University, Greenville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The West Clinic - Wolf River, Germantown, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (5):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No